CLINICAL TRIAL: NCT04306822
Title: Epidemiology of Cardiovascular Diseases and Their Risk Factors in Regions of Russian Federation
Acronym: ECVD-RF
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Collaborators: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government); Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 01201178178
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Risk Factor, Cardiovascular; Non-communicable Diseases; Cardiovascular Diseases
Keywords: epidemiology; risk factor; adult; non-communicable diseases; cardio-vascular diseases; dietary habits; arterial hypertension; smoking; physical activity; hypercholesterinemia
MeSH Terms: conditions — Noncommunicable Diseases; Cardiovascular Diseases; Feeding Behavior; Hypertension; Smoking; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study carried out in 2012-2014 years. The aim was to evaluate the prevalence of CVD and their RF in different regions of the Russian Federation and to develop epidemiological models of the CVD risk profile for the population based on traditional factors, as well as to assess the contribution of traditional and "new" cardiovascular risk factors to the mortality rate of the country's population based on domestic data. Thirteen regions were included. We examined 22,906 males and females, aged 25-64 years. The examination consist of anthropometry; the measurement of BP, resting heart rate, and a 12-lead standard electrocardiography (ECG) in a supine position. The personal interview information was collected using a structured questionnaire, and included socio-demographic and socio-economic measures; health parameters; medical history; stress, and depression. Continued monitoring of mortality, the latest mortality update includes deaths through 2019.

DETAILED DESCRIPTION:
The representative (systematic stratified multistage) random sample was generated according to the territorial principle (Kish method) in 13 regions of the Russian Federation. The study sample included 22,906 participants (8353 males and 13553 females) 25-64 years old, with a response rate - 80%, examined in 2012-2014. The following regions were included: Volgograd, Voronezh, Vologda, Ivanovo, Kemerovo, Orenburg, Samara, Tomsk, Tyumen regions, St. Petersburg, Krasnoyarsk, Primorsky Territory and the Republic of North Ossetia-Alania. All of the subjects were examined using a standard questionnaire consisting of 12 modules and containing information on age and gender composition, educational status, professional affiliation, level of well-being of survey participants, the presence of behavioral risk factors: smoking, excessive alcohol consumption, low physical activity, poor nutrition, as well as anxiety and depressive disorders. In addition, the questionnaire included anamnestic data on chronic diseases and drug therapy. Quality of life was assessed using the EUROQOL international questionnaire - EQ-5D All subjects were measured blood pressure (BP) and heart rate twice according to the standard procedure. Anthropometric procedures included measuring weight (kg), height (m), waist circumference (cm), calculating body mass index (BMI; kg / m2). The lipid profile was determined for all patients, including levels of HDL and HDL cholesterol, triglycerides, as well as glucose, creatinine and uric acid. The levels of these parameters in blood serum were determined by Abbot Architect c8000 biochemical analyzer (USA). The Additional Screening program, included sphygmomanometry, duplex scanning of carotid arteries, and evaluation of the parameters characterizing the functioning of metabolic systems (apo B and apo AI, as well as LP (a), C-reactive protein (hsCRP), NT-proBNP - the N-terminal propeptide of cerebral natriuretic hormone B-type, dash Nootropic hormone (TSH), insulin, D-dimer) in addition to the main survey was conducted in the 5 regions.Continued monitoring of mortality. Deaths were verified in residential registers and from telephone calls. The latest mortality update includes deaths through 2019.

ELIGIBILITY:
Inclusion Criteria:

* randomly selected males and females aged 25-64 years from 13 regions of Russian Federation

Exclusion Criteria:

* males and females younger than 24 years and older than 64 years

Ages: 25 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: The study participants were randomly selected from 13 regions of Russian Federation between 2012-2014. The final sample included 22,906 individuals (8353 males, 13553 females) who completed an interview and medical tests (response rate 80%).
Sampling Method: Probability Sample
Enrollment: 22906 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The number of fatal and non-fatal events | 6 years
  cardiovascular death, noncardiovascular death, all-cause death, the triple composite of cardiovascular death, non-fatal MI or non-fatal stroke, fatal MI, fatal stroke, non-fatal MI, non-fatal stroke, hospitalization for HF, coronary angiography, PCI, and CABG